CLINICAL TRIAL: NCT04004806
Title: Tracking Device Guided Feedback to Enhance Patient Physician Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Accreditation Council for Graduate Medical Education (Other)
Responsible Party: Principal Investigator, Andrei Brateanu, MD, Internal Medicine Residency Associate Program Director, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-782
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Physician Patient Relation; Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Intervention (No Intervention): Phase 1 (Observational phase): All residents and staff physicians rotating through the inpatient medicine services during the first three (3) months, who agreed to be a part of the study, will be provided with Hill Rom tracking devices to quantify the time spent at the patient's bedside by each member as part of the daily practice.
- Intervention (Experimental): Phase 2 (Intervention phase): The interventional phase will be six (6) months duration. During this period, the recorded time spent by the individual study participants at the patient's bedside will be compared to their respective peers, and percentile scores will be generated. Based on these percentile scores, the study participants will receive emails notifying them of the results. Participants whose scores fall in the lower 50th percentile will be encouraged to increase patient interaction times. Participants with scores in the top 50th percentile will receive congratulatory emails to encourage them to keep up the performance.
  Interventions: Device: Hill Rom tracking device
- Post-Intervention (No Intervention): Phase 3: (Post Intervention observation phase): The final phase of the study will be again three (3) months. The intervention of feedback emails and text pages will be discontinued and the study participants will only be monitored to see if the past intervention made an impact on their daily clinical practice in terms of time spent with the patients.

INTERVENTIONS:
Device: Hill Rom tracking device — Location tracking devices from Hill Rom company.
  Other Names: Feedback emails and text pages
  Arms: Intervention

SUMMARY:
A prospective cohort study aimed to determine the impact of increased physician patient interaction on physician well being and patient satisfaction. It involves recording time spent by physicians at the patient's bedside using tracking devices and providing feedback emails encouraging them to spend more time. The data will be analyzed to see if bedside time correlates with patient satisfaction scores.

The study has 3 phases - 1. Observational phase for 3 months: Only involves recording baseline physician bedside time using tracking devices. 2. Interventional phase for 6 months involves generating percentile scores for physician bedside time and providing feedback through emails and texts. 3. Post intervention phase for 3 months to evaluate the impact of intervention on daily practice of physicians.

DETAILED DESCRIPTION:
All residents and staff members who do not opt out of the study by July 1, 2019 will be included as the final study population. The planned duration of the study is 12 months starting from July 2019 - June 2020. The total time period will be further divided into three phases.

Phase 1 (Observational phase): All residents and staff physicians rotating through the inpatient medicine services during the initial 3 months who agreed to be a part of the study will be provided with Hill Rom tracking devices to quantify the time spent at the patient's bedside by each member as part of the daily practice.

Phase 2 (Intervention phase): Following the initial observational phase, the interventional phase will be 6 months in duration . During this period, the recorded time spent by the individual study participants at the patient's bedside will be compared to their respective peers (e.g. intern to intern, senior resident to senior resident and staff physician to staff physician), and percentile scores will be generated. Time spent by each member of each team at the patient's bedside will be abstracted from the tracking software daily and added on a weekly basis to generate cumulative values by the research coordinator. Patients not assigned to a particular team member will not count towards the denominator. Data will be collected individually for the staff physician, senior resident and intern in each team and compared to peer members in the other teams and converted to percentiles. Based on these percentile scores, the study participants will receive emails and text pages notifying them of the results. The participants whose scores fall in the lower 50th percentile, will be encouraged to increase patient interaction times to reach a target of at least 50th percentile. Striving to stay in the top 50th percentile will provide continuous reinforcement. The participants with scores in the top 50th percentile will receive congratulatory emails to encourage them to keep up the performance. In case of scheduling changes or absences, team members can notify the study coordinator to exclude their data for the said number of days. The percentile scores will be used solely for the purpose of this study and will neither impact trainee evaluation nor their learning objectives for the rotation. Similarly for staff physicians, the scores generated will not be a part of their annual performance reviews.

Phase 3: (Post Intervention observation phase): The final phase of the study will be 3 months. The intervention of feedback emails and text pages will be discontinued and the study participants will only be monitored to see if the past intervention made an impact on their daily clinical practice in terms of time spent with the patients.

At the end of the rotation the study participants will be assessed for their well-being and burnout by surveying them using the standard, validated, IRB-approved, anonymous questionnaires provided by the Accreditation Council for Graduate Medical Education (ACGME), during each of the above phases

ELIGIBILITY:
Inclusion Criteria:

* Cleveland Clinic Main Campus Internal Medicine resident or staff physician

Exclusion Criteria:

* Below the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Time spent at bedside | through study completion, one year
  total number of minutes spent by each participant at a patient's bedside divided by the total number of patients

SECONDARY OUTCOMES:
Physician burnout scores | through study completion, one year
  correlation of time spent by residents and physicians at the patient's bedside with their burnout survey results as measured by a questionnaire provided by the Accreditation Council for Graduate Medical Education (AGME) which consists of 22 fixed response and Likert-type scale questions.
HCAHPS Patient satisfaction scores | through study completion, one year
  correlation of time spent by residents and physicians at the patient's bedside with patient satisfaction scores as measured by HCAHPS v13 (based on question 5, 6 and 7 which form the 'Your Care from Doctors' section in the HCAHPS v 13.0, 2018 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Brateanu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States